CLINICAL TRIAL: NCT03132571
Title: A Pilot Trial of Naltrexone-Bupropion Combination Versus Placebo Combined With Bupropion for Weight Loss in Comorbid Schizophrenia
Brief Title: Naltrexone-Bupropion Versus Placebo-Bupropion for Weight Loss in Schizophrenia
Acronym: NBC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued due to funding.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1606017928
Record Dates: First submitted 2017-04-17; First posted 2017-04-28 (Actual); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Diabetes Mellitus, Type 2; Obesity
Keywords: Schizophrenia; Diabetes; Obesity
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Naltrexone; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Naltrexone versus Placebo assignment will remain double-blinded for the duration of the study; Bupropion dosing will be open-label and not masked to either participant or investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone with Bupropion (Experimental): Oral Naltrexone taken once a day and Oral Bupropion taken once a day for 16 weeks.
  Interventions: Drug: Naltrexone; Drug: Bupropion
- Placebo with Bupropion (Placebo Comparator): Oral placebo capsule and Oral Bupropion taken once a day for 16 weeks.
  Interventions: Drug: Bupropion; Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — 37.mg oral capsule taken once daily for over the course of the study (16 weeks)
  Other Names: Revia
  Arms: Naltrexone with Bupropion
Drug: Bupropion — Extended release bupropion taken once daily for the course of the study (16 weeks) flexible dosing up to 450mg target.
  Other Names: Wellbutrin; Zyban
Other: Placebo — Oral placebo taken once daily for the course of the study (16 week)
  Arms: Placebo with Bupropion

SUMMARY:
The purpose of this study is to determine the efficacy of combining open-label extended release bupropion (flexible dosing up to 450mg target) and naltrexone (37.5mg) versus Bupropion and placebo along with a daily 500 calorie reduction diet recommendation for weight and health risk reduction in 40 overweight/obese individuals with schizophrenia.

DETAILED DESCRIPTION:
The combination of naltrexone with noradrenaline/dopamine reuptake blocker bupropion has been developed and FDA-approved for the treatment of obesity in the general population. Naltrexone does not normally produce weight loss in humans and bupropion produces modest weight loss, however the combination produces clinically significant weight loss, which appears to be more than the sum of its components would otherwise produce separately. Of interest to us, the combination has been shown to be effective for clinically significant weight loss in obese subjects with type 2 diabetes as well. Registration studies by the manufacturer of the combination pill excluded antipsychotic medication users, thus we have no information on the potential effectiveness of the combination in this population. Both naltrexone and bupropion are commonly used in psychiatry, naltrexone for co-morbid alcohol addiction, and bupropion for co-morbid depression and/or cigarette addiction. This is a 16-week pilot trial of 37.5mg naltrexone/placebo added to extended release bupropion in flexible dosing (150mg to 450mg) and a daily 500 calorie reduction diet recommendation for subjects with schizophrenia and obesity. A dose of 37.5mg is similar to the FDA-approved combination dose for naltrexone. However, based on our experience with bupropion, we have chosen to use bupropion in an un-blinded manner and reach the target dose of 450mg based on tolerance of the individual subject over the initial 3-week period.

Changes to the study since registration:

The study was initially registered with 3 arms (Naltrexone vs Bupropion vs Placebo)- whereas the original intent was always supposed to be a 2 armed study (Naltrexone vs Placebo- each with Bupropion included)- this was corrected when the results of the terminated study were entered. In addition, there was an initial intent to include diabetics in the study, but this was later removed as well.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 to 75
2. Meet DSM-IV criteria for schizophrenia or schizoaffective disorder based on SCID interview (If bipolar-schizoaffective: need to be adequately stabilized on a mood stabilizer and show no mania history for the past one year, as confirmed by study psychiatrist and patient's clinician)
3. Body Mass Index (BMI) of 28 and over
4. On a stable dose of antipsychotic medication; i.e. at least one month with no dose change, and three months from an antipsychotic switch
5. Deemed to be symptomatically stable by the clinical staff in the last two months
6. Over 7% total body weight increase on antipsychotics for subjects within first year of illness

Exclusion Criteria

1. Meet criteria for current opiate abuse or dependence (confirmed by positive urine drug screen for opiates or, if suspected by study doctor via patient history and or suspicion of occult opiate use.) Note: All subjects will be screened for drugs, not only those suspected of opiate use.
2. A history of seizures in the past five years (confirmed through chart review and discussion with patient's clinician)
3. Meet DSM criteria for Bipolar Disorder
4. History of mania in the past one year (confirmed through chart review and discussion with patient's clinician)
5. Uncontrolled hypertension
6. Insulin dependent diabetes mellitus
7. Current history of dementia, mental retardation
8. Not capable of giving informed consent for participation in the study
9. Women who are pregnant or breast-feeding
10. Physical conditions affecting body weight (e.g. Cushing's disease, polycystic ovary syndrome)
11. Severe liver dysfunction, (serum aminotransferases greater than three times normal), acute infectious hepatitis, liver failure.
12. History of glaucoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data resulting from this award involving human subjects will be submitted to the NIMH Data Archive (NDA) - National Database for Clinical Trials Related to Mental Illness (NDCT) The Principal Investigator will work with NDA support staff to plan an appropriate data submission schedule and provide information on the steps for submission and sharing of data. Communication of this data sharing plan to appropriate research staff to ensure the timely submission of data. All human subject data provided will include an NDA Global Unique Identifier (GUID) and will not include personally identifiable information (PII). Analyzed data will be submitted no later than the time of publication. Even if a publication focuses on only part of an analyzed dataset, the entire analyzed dataset will be submitted when the first paper is published. All data made available for public use via NDA will be de-identified data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 people were screened by telephone.
  18/30 people screened were deemed ineligible. The reasons for ineligibility were: antidepressant medication use (11/18), a history of seizures (4/18) and already taking Naltrexone (3/18).
  12/30 people were eligible, 6/12 were initially interested in the study and ultimately, only 5/6 were consented.
Period: Overall Study
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.33 (8.14) | 58.00 (1.41) | 51.00 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: BMI
Description: BMI will be calculated using weekly height and weight measurements (kg/m^2) at each assessment.
Time Frame: Baseline and Week 16
Population: Presented are the baseline and 16 weeks summary data on the 5 patients enrolled.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
Number analyzed (Participants) | 3 | 2
kg/m^2
  Baseline | 39.06 (6.03) | 29.55 (0.07)
  16 Weeks | 37.33 (5.81) | 30.65 (3.88)

2. Secondary Outcome: Weight (kg)
Description: Weight in kilograms will be measured at each assessment and change will be determined at study endpoint.
Time Frame: Baseline and Week 16
Population: Presented are the baseline and 16 weeks summary data on the 5 patients enrolled.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
Number analyzed (Participants) | 3 | 2
kg
  Baseline | 118.78 (11.17) | 87.25 (15.48)
  16 Weeks | 113.60 (11.24) | 91.25 (27.64)

3. Secondary Outcome: Health Risk Markers
Description: Serum lipid profiles, fasting glucose, and glycosylated hemoglobin (hbA1c) will be measured at baseline and week 16 and change in these markers will be determined at endpoint
Time Frame: Baseline to Week 16
Population: These labratory data were not collected and summarized due to the removal of diabetes from the study criteria and the early termination of the study.
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Waist Circumference (Inches)
Description: Waist circumference will be measured in inches at each assessment.
Time Frame: Baseline and Week 16
Population: Presented are the baseline and 16 weeks summary data on the 5 patients enrolled.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
Number analyzed (Participants) | 3 | 2
inches
  Baseline | 50.08 (5.26) | 41.87 (1.23)
  16 Weeks | 48.50 (5.76) | 43.37 (2.29)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored in patients up to 16 weeks post randomization.
Arm/Group | Naltrexone With Bupropion | Placebo With Bupropion
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone With Bupropion (N=3) | Placebo With Bupropion (N=2)
Nausea (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT03132571/Prot_SAP_000.pdf